CLINICAL TRIAL: NCT03574571
Title: Phase III Trial of Docetaxel vs. Docetaxel and Radium-223 for Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: A Study to Test Radium-223 With Docetaxel in Patients With Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-150; 2018-002944-10 (EudraCT Number)
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Radium-223; Docetaxel; 18-150; C16-174; DORA Trial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Radium-223

STUDY DESIGN:
Intervention Model Description: This is an open-labeled, randomized, phase III study of docetaxel versus docetaxel in combination with radium-223 in subjects with mCRPC.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel (Experimental): Docetaxel 75 mg/m2 will be administered IV every three weeks for 10 doses. Prednisone will be given at a dose of 5mg orally twice daily.
  Interventions: Drug: Docetaxel 75 mg/m2
- Docetaxel with Radium-223 (Experimental): Docetaxel 60 mg/m2 will be administered IV every 3 weeks for 10 doses. Radium-223 will be administered at 55 kBq/kg, 6 injections at 6 weeks intervals.
  Interventions: Drug: Docetaxel 60 mg/m2; Drug: Radium-223

INTERVENTIONS:
Drug: Docetaxel 75 mg/m2 — Docetaxel 75 mg/m2 will be administered IV every three weeks for 10 doses.
  Arms: Docetaxel
Drug: Docetaxel 60 mg/m2 — Docetaxel 60 mg/m2 will be administered IV every 3 weeks for 10 doses.
  Arms: Docetaxel with Radium-223
Drug: Radium-223 — Radium-223 will be administered at 55 kBq/kg, 6 injections at 6 weeks intervals.
  Arms: Docetaxel with Radium-223

SUMMARY:
The purpose of this study is to compare any good and bad effects of using radium-223 along with docetaxel chemotherapy treatment versus using docetaxel alone. Earlier studies helped show that the combination is safe, but the combination has not been proven to work better than either drug alone. The goal of this study is to find out if combining docetaxel and radium-223 is better than giving either drug by itself.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent (ICF) and HIPAA authorization for the release of personal health information. A signed informed consent must be obtained before screening procedures are performed.

NOTE: HIPAA authorization may be either included in the informed consent or obtained separately.

* Males 18 years of age and above
* Histological or cytological proof of prostate cancer
* Documented progressive mCRPC based on at least one of the following criteria:

  1. PSA progression defined as 25% increase over baseline value with an increase in the absolute value of at least 1.0 ng/mL that is confirmed by another PSA level with a minimum of a 1 week interval and a minimum PSA of 1.0 ng/mL.
  2. Soft-tissue progression defined as an increase ≥ 20% in the sum of the LD of all target lesions based on the smallest sum LD since treatment started or the appearance of one or more new lesions.
  3. Progression of bone disease (evaluable disease) or two or more new bone lesions by bone scan.
* Two or more bone lesions
* ECOG 0- 1
* Normal organ function with acceptable initial laboratory values within 14 days of randomization:

  * Albumin > 30 g/L
  * ANC ≥ 1.5 x 10^9/L
  * Hemoglobin ≥ 10 g/dL
  * Platelet count ≥ 100 x 10^9/L
  * Creatinine ≤ 1.5 x the institutional upper limit of normal (ULN)
  * Bilirubin ≤ ULN (unless documented Gilbert's disease)
  * SGOT (AST) ≤ 1.5 x ULN
  * SGPT (ALT) ≤ 1.5 x ULN
  * WBC count ≥ 3 x 10^9/L
* Subjects must agree to use a medically acceptable method of birth control (e.g., spermicide in conjunction with a barrier such as a condom) or sexual abstinence for the duration of the study, including 30 days after the last dose of study drug. Sperm donation is prohibited during the study and for 30 days after the last dose of study drug. Female partners must use hormonal or barrier contraception unless postmenopausal or abstinent.
* Serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH analogue (agonist or antagonist) if they have not undergone orchiectomy.
* All acute toxic effects of any prior treatment have resolved to NCI-CTCAE v4.0 Grade 1 or less.
* Willing and able to comply with the protocol, including follow-up visits and examinations

Exclusion Criteria:

* Received any other investigational therapeutic agents or other anticancer therapies within 4 weeks prior to randomization.

  °Note: If this requirement to have a washout of 2 weeks or 5 half-lives prior to randomization causes potential treatment delay due to Radium-223 importation timelines, the PCCTC must be contacted at pcctc@mskcc.org to request approval to randomize the subject prior to the completion of the washout. Requests for early randomization must be accompanied by written assurance by the site that the washout will be completed prior to treatment start.
* Received external beam radiotherapy within the 4 weeks prior to randomization.

  ° Note: If prolonging randomization to complete EBRT washout causes potential treatment delay due to Radium-223 importation timelines, the PCCTC must be contacted at pcctc@mskcc.org to request approval to randomize the subject prior to the completion of the washout. Requests for early randomization must be accompanied by written assurance by the site that the washout will be completed prior to treatment start.
* Has an immediate need for external beam radiotherapy.
* Has received any systemic bone-seeking radiopharmaceutical in the past.
* Has received any prostate cancer directed chemotherapy in the castration resistant setting. Subjects who have received up to 6 prior doses of docetaxel in the castration sensitive setting are permitted if they have not experienced disease progression within 36 weeks of last treatment with docetaxel.
* Has received four or more systemic anticancer regimens for mCRPC.

  * Treatment with docetaxel or abiraterone for non-castrate metastatic disease is permissible and does not count towards the lines of therapy for mCRPC
  * A 'line' is a regimen. Combinations of hormones and other types of therapies count as single lines.
* Has known Grade ≥3 docetaxel-related toxicities or docetaxel toxicity related dose interruption or discontinuation.
* Has received blood transfusions or growth factors within the last 4 weeks prior to randomization.
* Symptomatic nodal disease (i.e., scrotal, penile, or leg edema).
* Has visceral metastases with ≥ 3 lung and/or liver metastases or individual lesion ≥2 cm, as assessed by CT scan or MRI of the chest/abdomen/pelvis within the last 8 weeks prior to randomization.
* Symptomatic loco-regional disease that causes ongoing Grade 3 or Grade 4 urinary or rectal symptoms.
* Subjects with a "currently active" second malignancy other than non-melanoma skin cancers or non-invasive bladder cancers or other in-situ or non-invasive malignancies. Subjects are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years.
* Has imminent or established cord compression based on clinical findings and/or MRI.
* Known bone marrow dysplasia
* Has received any of the following in the 4 weeks prior to randomization: 5-alpha-reductase inhibitors, herbal medications, natural hormonally active foods (e.g., phytoestrogens) or other food supplements known to alter PSA in humans
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous, including but not limited to:

  * Uncontrolled infection
  * NYHA III or IV heart failure
  * Crohn's disease or those with ulcerative colitis who have not undergone a colectomy
  * Known active infection with HIV, Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate
Enrollment: 732 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival is defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (72):
- United States (40):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Yale University- Yale Cancer Center, New Haven, Connecticut
  - Helen Graham Cancer Center (Christiana Care), Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Mount Sinai Medical Center (Miami), Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - New Jersey Urology, Saddle Brook, New Jersey
  - New Mexico Oncology and Hematology, Albuquerque, New Mexico
  - University of Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York
  - Bronx VA Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health/ Levine Cancer Institute, Monroe, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Dayton Physicians Network, Kettering, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Research Institute, Houston, Texas
  - Millennium Physicians, Houston, Texas
  - University of Washington, Seattle, Washington
- Brazil (10):
  - Hospital de Amor de Barretos (Fundação Pio XII) / Barretos Cancer Hospital, Barretos, Dr. Paulo Prata
  - Instituto de Medicina Integral Professor Fernando Figueira (IMIP), Boa Vista, Pernambuco
  - Instituto Brasileiro de Controle do Câncer/IBCC, São Paulo, State of São Paulo
  - Hospital Sírio Libanês, Brasília
  - Hospital Erasto Gaertner, Curitiba
  - CPORS - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre
  - Hospital Moinhos de Vento (HMV), Porto Alegre
  - Hospital Israelita Albert Einstein, São Paulo
  - Beneficência Portuguesa, São Paulo
  - Centro de Pesquisas São Lucas - Sociedade Campineira de Educação e Instrução (SCEI), São Paulo
- Netherlands (13):
  - Nederlands Kanker Instituut, Amsterdam, Plesmanlaan
  - Noordwest Ziekenhuisgrouep Alkmaar (NWZ), Alkmaar
  - Ziekenhuisgroep Twente (ZGT), Almelo
  - Amphia Hospital, Breda
  - Deventer Ziekenhuis, Deventer
  - Tergooi Hospital, Hilversum
  - Canisius Wilhelmina Ziekenhuis (CWZ), Nijmegen
  - Erasmus MC Cancer Institute, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Maasstad Hospital, Rotterdam
  - Haaglanden Medical Center, The Hague
  - St. Antonius Ziekenhuis (Utrecht), Utrecht
  - Isala Kliniek, Zwolle
- Spain (9):
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Avenida de Roma S/n
  - Ramón y Cajal Hospital, Madrid, Madrid
  - Hospital Del Mar, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - Clinic de Barcelona, Barcelona
  - Hospital Provincial de Castellón, Castellon
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm